CLINICAL TRIAL: NCT00719511
Title: Single Center Phase I/IIa, Placebo Controlled, Randomized, Double-blind, Dose-response Study to Assess the Optimal Dose as Well as Clinical Efficacy and Safety of a Novel Method of Specific Allergen Immunotherapy in Grass Pollen Allergic Subjects by Epicutaneous Allergen Administration
Brief Title: Study of Specific Allergen Immunotherapy in Grass Pollen Allergic Subjects by Epicutaneous Allergen Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: PD Dr. Thomas Kündig, University Hospital Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZU-SkinSIT-002
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Allergies
Keywords: Rhinoconjunctivitis; Allergic
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Patch allergen dose 1
  Interventions: Drug: Purified allergen dose 1 integrated in a Patch system
- 2 (Experimental): Patch allergen dose 2
  Interventions: Drug: Purified allergen dose 2 integrated in a Patch system
- 3 (Experimental): Patch allergen dose 3
  Interventions: Drug: Purified allergen dose 3 integrated in a Patch system
- 4 (Experimental): Placebo
  Interventions: Drug: Purified allergen integrated in a Patch system

INTERVENTIONS:
Drug: Purified allergen dose 1 integrated in a Patch system — Epicutaneous application of a patch
  Arms: 1
Drug: Purified allergen dose 2 integrated in a Patch system — Epicutaneous application of a patch
  Arms: 2
Drug: Purified allergen dose 3 integrated in a Patch system — Epicutaneous application of a patch
  Arms: 3
Drug: Purified allergen integrated in a Patch system — Epicutaneous application of a patch
  Arms: 4

SUMMARY:
Evaluation of patch as specific immunotherapy in allergic patients

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* History of grass pollen allergic rhinitis
* Male and female between 18 years to 65 years
* Positive skin-prick test to grass pollen
* Positive conjunctival provocation test

Exclusion criteria:

* Eczematous skin lesions on the upper arms
* Perennial allergic rhinitis
* Symptoms of infectious disease with rhinitis in between the last 2 weeks
* Surgical intervention in between the last 30 days
* Pregnancy or nursing
* History of HIV or AIDS
* History of mastocytosis (cutaneous or systemic)
* History of significant cardiovascular disease
* Hypertension (blood pressure > 160 / 95)
* History of significant pulmonary, renal and/or hepatic disease
* History of significant hematological disorder
* Moderate or severe asthma
* History of malignancy
* History of neurological or psychiatric disease
* History of autoimmune disease
* Antihistamines with longed half-lives in the last week
* Systemic or topical steroids for 5 days
* Active infectious disease
* Contraindicated medications:

  * immunosuppressive agents
  * Betablockers
  * ACE-inhibitors, AT 2 Antagonists
  * tricyclic antidepressants
  * daily use of Beta-agonists or steroid inhalers
* Participation in another clinical trial /study at the moment or within the last 60 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of the placebo with that of three different test doses of the epicutaneous pollen allergen administration evaluated by visual analog scales after the treatment | 2010

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland